CLINICAL TRIAL: NCT02869919
Title: Vitamin D Levels in Critically Ill Patients With Acute Kidney Injury
Brief Title: Vitamin D in Critically Ill Patients With Acute Kidney Injury
Acronym: VID-AKI
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 196968
Record Dates: First submitted 2016-05-16; First posted 2016-08-17 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with AKI: critically ill patients with acute kidney injury
  Interventions: Other: AKI
- Patients without AKI: critically ill patients without acute kidney injury
  Interventions: Other: AKI

INTERVENTIONS:
Other: AKI — Vitamin D levels

SUMMARY:
This study aims to investigate whether there is a difference in Vitamin D levels between critically ill adult patients with and without acute kidney injury.

DETAILED DESCRIPTION:
Vitamin D has an important role in calcium homeostasis and the regulation of bone metabolism. It also appears to play a role in various infectious, immunologic, neurologic, cardiovascular and respiratory disorders. Both, biological and observational studies have identified vitamin D deficiency as a risk factor for adverse outcomes during critical illness. However, administration of high dose vitamin D to a general population of critically ill patients with vitamin D deficiency did not reduce mortality or hospital length of stay. The exception was a pre-defined sub-group of patients with Vitamin D levels in the very low range (<30 nmol/L) where hospital mortality was significantly lower in patients treated with Vitamin D.

Vitamin D Metabolism The majority of vitamin D is produced through the direct action of sunlight on 7-dehydrocholesterol in the skin. The inert Vitamin D3 produced in this manner, together with Vitamin D2 or D3 from dietary sources, require hydroxylation in the liver to 25-hydroxyvitamin D [25(OH)D] which is the main circulating form. Conversion of this still inactive substance to the active form, 1,25-dihydroxyvitamin D [1,25(OH)2D], by the enzyme 1α-hydroxylase occurs primarily, but not exclusively, in the proximal renal tubules. Circulatory phosphorous, parathyroid hormone (PTH) and fibroblast growth factor 23 (FGF23) play an important regulatory role in this process. FGF23 is a bone derived hormone that inhibits renal tubular absorption of phosphate and reduces circulating 1,25(OH)2D. PTH is a hormone secreted by the parathyroid glands in response to hypocalcaemia. It acts to increase the concentration of calcium through several pathways one of which is the upregulation of 1α-hydroxylase, the enzyme responsible for converting 25(OH)D to 1,25(OH)2D.

The majority of both 25(OH)D and 1,25(OH)2D is bound to Vitamin D Binding Protein (VDBP) in circulation. The nuclear Vitamin D Receptors (VDR) which regulate the transcription and expression of Vitamin D targeted genes are only activated by unbound 1,25(OH)2D, which is less than 1% of total circulating Vitamin D.

Vitamin D in chronic kidney disease In patients with chronic kidney disease (CKD) on chronic dialysis, Vitamin D deficiency is common (>80%), and the supplementation with active Vitamin D preparations is strongly recommended to prevent or ameliorate the effects of hyperparathyroid high-turnover bone disease and to reduce the cardiovascular risk.

Vitamin D in general ICU patients ICUs worldwide have reported Vitamin D deficiency ranging from 60-100%. A randomized controlled trial (RCT) in a general population of critically ill patients with vitamin D deficiency showed that administration of high dose vitamin D did not reduce mortality or hospital length of stay. The exception was a pre-defined sub-group of patients with Vitamin D levels in the very low range (<30 nmol/L) in whom hospital mortality was significantly lower in patients treated with Vitamin D. Another RCT investigated the role of 2 different doses of cholecalciferol in 50 critically ill adults with the systemic inflammatory response syndrome. The study showed that prior to randomization 56% of patients were classified as Vitamin D deficient. By day 7 after randomization, Vitamin D levels normalized in >60% of patients and PTH levels decreased over the study period.

Vitamin D and AKI AKI is an abrupt deterioration in kidney function which develops over hours or days for a variety of reasons and can range from mild impairment to acute kidney failure. It affects >50% of critically ill patients worldwide and is independently associated with an increased risk of complications, a longer stay in hospital and high risk of dying. AKI survivors have an increased risk of CKD and premature mortality. A recent study also confirmed a significantly increased risk of bone fractures in patients who survived an episode of AKI requiring renal replacement therapy (RRT).

The causal mechanisms behind the morbidity and mortality associated with AKI are still not fully understood but Vitamin D may play an important role.

The hypothesis of this study is that critically ill patients with AKI have significantly lower Vitamin D levels than critically ill patients without AKI.

ELIGIBILITY:
Inclusion Criteria:

age >18 years presence of organ failure

Exclusion Criteria:

Chronic kidney disease stage 3b-5 Renal Transplant Vitamin D deficiency Vitamin D supplementation Hyperparathyroidism Treatment with total parenteral nutrition Life expectancy <48 hours Patients with haemoglobin <70g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients in the Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | up to 28 days

SECONDARY OUTCOMES:
PTH levels | up to 28 days
FGF23 levels | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, PhD, Principal Investigator — Guy's & St Thomas Hospital
Locations (1):
- Guy's & St Thomas Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No We are not planning to make individual participant data available

REFERENCES:
- [Derived] Cameron LK, Ledwaba-Chapman L, Voong K, Hampson G, Forni LG, Seylanova N, Harrington DJ, Lim R, Bociek A, Yanzhong W, Ostermann M. Vitamin D metabolism in critically ill patients with acute kidney injury: a prospective observational study. Crit Care. 2024 Apr 2;28(1):108. doi: 10.1186/s13054-024-04869-4. PMID 38566240
- [Derived] Cameron LK, Lei K, Smith S, Doyle NL, Doyle JF, Flynn K, Purchase N, Smith J, Chan K, Kamara F, Kidane NG, Forni LG, Harrington D, Hampson G, Ostermann M. Vitamin D levels in critically ill patients with acute kidney injury: a protocol for a prospective cohort study (VID-AKI). BMJ Open. 2017 Jul 12;7(7):e016486. doi: 10.1136/bmjopen-2017-016486. PMID 28706103